CLINICAL TRIAL: NCT02599961
Title: An Open-label Extension Study to Assess the Long-term Safety and Efficacy of UX007 in Subjects With Glucose Transporter Type 1 Deficiency Syndrome
Brief Title: Study to Assess the Long Term Safety and Efficacy of UX007 in Participants With Glucose Type 1 Deficiency Syndrome (Glut1 DS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was halted prematurely due to lack of efficacy
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX007G-CL202; 2015-000389-69 (EudraCT Number)
Expanded Access: NCT03773770 (Available)
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Results first posted 2020-04-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Glucose Transporter Type 1 Deficiency Syndrome
Keywords: Glut 1 DS
MeSH Terms: conditions — Glut1 Deficiency Syndrome | interventions — triheptanoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UX007 (Experimental): UX007 dosing targeted and/or maintained at 35% of total daily caloric intake.
  Interventions: Drug: UX007

INTERVENTIONS:
Drug: UX007 — UX007 is a liquid intended for oral (PO) administration.
  Other Names: Triheptanoin

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of UX007 in Glut1 DS participants.

DETAILED DESCRIPTION:
The study will enroll up to 40 pediatric, adolescent and adult Glut 1 DS participants who have completed the UX007G-CL201 (NCT019933186) study and, at the discretion of the Sponsor, additional participants from other clinical studies, investigator sponsored trials (ISTs), or expanded access/compassionate use treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Glut 1 DS confirmed by cerebrospinal fluid glucose concentration. erythrocyte 3-O-methyl-D-glucose uptake assay, or solute carrier family 2 member 1 (SLC2A1) molecular genetic testing (Information obtained from Medical Records)
* Males and females aged at least 1 year old at the time of informed consent
* Completion of UX007G-CL201 study (NCT01993186). Glut1 DS patients who received UX007/triheptanoin treatment as apart of clinical studies, ISTs or expanded access/compassionate use treatment programs may be eligible at the discretion of the Sponsor
* Provide written informed consent or verbal assent (if possible) with written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research related procedures
* Must, in the opinion of the investigator, be willing and able to complete all aspects of the study, and comply with accurate completion of the seizure diary
* Females of childbearing potential must have a negative urine pregnancy test at Baseline and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have not experienced menarche, are post-menopausal (defined as having no menses for at least 12 months without an alternative medical cause), or are permanently sterile due to total hysterectomy, bilateral salpingectomy, or bilateral oophorectomy.
* Participants of child-bearing potential or fertile males with partners of child-bearing potential who are sexually active must consent to use a highly-effective method of contraception as determined by the investigator from the period following the signing of the informed consent through 30 days after last dose of study drug.

Exclusion Criteria:

* Any known hypersensitivity to triheptanoin, that in the judgement of the investigator, places the subject at an increased risk for adverse effects
* History of, or current suicidal ideation, behavior and/or attempts
* Pregnant and/or breast feeding an infant
* Unwilling or unable to discontinue use of prohibited medication (barbiturates, pancreatic lipase inhibitors) or other substance that may confound study objectives. Use of up to 3 concomitant antiepileptic drugs is allowed, provided dose has been stable at least 14 days prior to Baseline
* Use of any Investigational Product, drug or supplement (other than UX007) within 30 days prior to Baseline, or at any time during the study
* Has a condition of such severity and acuity, in the opinion of the investigator, that it warrants immediate surgical intervention or other treatment
* Has a concurrent disease or condition, or laboratory abnormality that, in the view of the investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or introduce additional safety concerns

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09-10 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (9):
- United States (5):
  - Children's Hospital Colorado - University of Colorado, Denver, School of Medicine, Aurora, Colorado
  - Miami Children's Hospital, Miami, Florida
  - Columbia University Medical Center, New York, New York
  - Cook Children's Medical Center, Fort Worth, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Melbourne Brain Centre, Heidelberg, Victoria, Australia
- Copenhagen University Hospital, Copenhagen, Denmark
- Hospital Sant Joan De Deu, Barcelona, Spain
- The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

REFERENCES:
- See also: Company Website — http://www.ultragenyx.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled pediatric, adolescent, and adult glucose transporter type 1 deficiency syndrome (Glut1 DS) participants who completed the UX007G-CL201 study (NCT01993186; rollover participants). No non-rollover participants (those from other clinical studies, investigator sponsored trials, or expanded access/compassionate use treatment) enrolled.
Pre-assignment Details: For continuing UX007G-CL201 participants, the Week 52 visit of that study may have been conducted in conjunction with the Baseline visit for this study to avoid duplication of assessments.
Groups:
- UX007 (Triheptanoin): UX007 dosing was targeted and/or maintained at 35% of total daily caloric intake.
Period: Overall Study
Arm/Group | UX007 (Triheptanoin)
Started | 15
Completed | 0
Not Completed | 15
Not completed — Withdrawal by Subject | 1
Not completed — Subject Non-Compliance | 2
Not completed — Discontinuation of Study by Sponsor | 9
Not completed — Other, Not Specified | 3

BASELINE CHARACTERISTICS:
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.24 (6.106)
Age, Customized [Count of Participants; unit: Participants]
  2 to < 12 years | 5
  12 to < 18 years | 5
  18 to < 65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Black or African American | 1
  White | 11
  Other, Not Specified | 1
Overall Seizure Frequency Per 4 Weeks [Mean (Standard Deviation); unit: seizures per 4 weeks] — The number of observable seizures were recorded by the subject or caregiver via diary. Observable seizures were defined as: generalized tonic-clonic; generalized tonic; generalized clonic; generalized atonic; partial/focal with secondary generalization; myoclonic, myoclonic (astatic) atonic, myoclonic tonic; complex partial/focal; simple partial/focal motor; absence.
  seizures per 4 weeks | 312.17 (528.057)
Baseline (NCT01993186) Columbia Neurological Score (CNS) Total Score [Mean (Standard Deviation); unit: score on a scale] — The CNS evaluates measures of neurological function and development delay, and is the sum of scores for the following domains: Weight, Height, Head Circumference, General Medical Exam, Funduscopic Exam, Cranial Nerves, Stance & Gait, Involuntary Movements, Sensation, Cerebellar Function, Muscle Bulk, Tone & Strength, Myotatic Reflexes, Toe Sign, Other Findings. The CNS is only scored when all domains are measured and ranges from 0 (abnormal exam) to 76 (normal exam). Higher scores are associated with higher neurological function. Population: participants with a baseline assessment
  score on a scale
    number analyzed (Participants) | 12
    (all) | 38.63 (25.428)
Baseline (NCT01993186) Short Form (SF) 10 (SF-10) Health Survey for Children Physical Summary Score [Mean (Standard Deviation); unit: T-score] — The SF-10 Health Survey for Children was administered to caregivers of participants aged 5-17 years. Responses are used to generate 2 component summary scores: Physical Summary Score and the Psychosocial Summary Score. The T-score based scale scores were centered so that a score of 50 corresponds to the average score in a comprehensive 2006 sample (a combination of general population and supplemental disability and chronic condition samples). Higher scores are associated with better quality of life. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 10
    (all) | 32.63 (17.027)
Baseline (NCT01993186) SF-10 Health Survey for Children Psychosocial Summary Score [Mean (Standard Deviation); unit: T-score] — The SF-10 Health Survey for Children was administered to caregivers of participants aged 5-17 years. Responses are used to generate 2 component summary scores: Physical Summary Score and the Psychosocial Summary Score. The T-score based scale scores were centered so that a score of 50 corresponds to the average score in a comprehensive 2006 sample (a combination of general population and supplemental disability and chronic condition samples). Higher scores are associated with better quality of life. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 10
    (all) | 48.29 (10.196)
Baseline (NCT01993186) SF12 Version 2 (SF-12v2) Health Survey Physical Component Summary (PCS) Score [Mean (Standard Deviation); unit: T-score] — SF-12v2 was assessed for adults aged >=18 years. Eight domain scores were used to generate 2 component summary scores: physical health (PCS) and mental health (MCS). The PCS and MCS scores have mean of 50 and SD of 10. The T-score based scoring method scores the data in relation to US general population T-scores. Therefore, all scores obtained that are < 50 can be interpreted as below the US general population T-score and scores > 50 can be interpreted as above the US general population T-score. Higher global scores are associated with better quality of life. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 2
    (all) | 39.37 (0.523)
Baseline (NCT01993186) SF-12v2 Health Survey MCS Score [Mean (Standard Deviation); unit: T-score] — SF-12v2 was assessed for adults aged >=18 years. Eight domain scores were used to generate 2 component summary scores: physical health (PCS) and mental health (MCS). The PCS and MCS scores have mean of 50 and SD of 10. The T-score based scoring method scores the data in relation to US general population T-scores. Therefore, all scores obtained that are < 50 can be interpreted as below the US general population T-score and scores > 50 can be interpreted as above the US general population T-score. Higher global scores are associated with better quality of life. Population: participants with a baseline assessment
  T-score
    number analyzed (Participants) | 2
    (all) | 43.49 (4.356)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Discontinuations Due to TEAEs, and Deaths
Description: An adverse event (AE) was defined as any untoward medical occurrence, whether or not considered drug related. Serious adverse events (SAEs) are AEs that at any dose, in the view of either the investigator or sponsor, results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or disability; a congenital anomaly/birth defect; other important medical event. An AE was considered a TEAE if it occurred on or after the first dose in this study, and was not present prior to the first dose in this study, or it was present at the first dose in this study but increased in severity during the study. Severity was based on Common Terminology Criteria for Adverse Events (CTCAE): 1 = mild, 2 = moderate, 3 = severe, 4 = life threatening, and 5 = death related to AE.
Time Frame: From first dose of study drug up to 36 months. The mean (SD) treatment duration was 667.9 (357) days.
Measure: Count of Participants; unit: Participants
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 15
Participants
  TEAEs | 13
  Serious TEAEs | 2
  Related TEAEs | 10
  Serious and Related TEAEs | 0
  Grade 3 or 4 TEAEs | 1
  Gastrointestinal TEAEs | 9
  TEAEs Leading to Treatment Discontinuation | 0
  TEAEs Leading to Study Discontinuation | 0
  TEAEs Leading to Death | 0

2. Secondary Outcome: Change From Baseline Over Time in Overall Seizure Frequency Per 4 Weeks
Description: The number of observable seizures were recorded by the subject or caregiver via diary throughout the study. Observable seizures were defined as: generalized tonic-clonic; generalized tonic; generalized clonic; generalized atonic; partial/focal with secondary generalization; myoclonic, myoclonic (astatic) atonic, myoclonic tonic; complex partial/focal; simple partial/focal motor; absence.
Time Frame: Baseline (from NCT01993186), Month 0-3, Month 4-6, Month 7-9, Month 10-12, Month 13-18, Month 19-24, Month 25-30, Month 31-36
Population: Participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: seizures per 4 weeks
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 15
seizures per 4 weeks
  Change at Month 0-3: number analyzed (Participants) | 10
  Change at Month 0-3 | -64.22 (185.564)
  Change at Month 4-6: number analyzed (Participants) | 7
  Change at Month 4-6 | -64.19 (142.460)
  Change at Month 7-9: number analyzed (Participants) | 7
  Change at Month 7-9 | -61.81 (164.770)
  Change at Month 10-12: number analyzed (Participants) | 7
  Change at Month 10-12 | -91.93 (216.834)
  Change at Month 13-18: number analyzed (Participants) | 8
  Change at Month 13-18 | -75.56 (206.406)
  Change at Month 19-24: number analyzed (Participants) | 6
  Change at Month 19-24 | -110.12 (233.492)
  Change at Month 25-30: number analyzed (Participants) | 5
  Change at Month 25-30 | -135.60 (249.871)
  Change at Month 31-36: number analyzed (Participants) | 2
  Change at Month 31-36 | -51.88 (101.378)
Statistical Analysis 1: Comparison: UX007 (Triheptanoin); Month 0-3; Test type: Superiority; p < 0.0001, generalized estimating equation (GEE) — From the GEE model which includes the reduction from baseline for each visit period as the response variable, baseline as covariates, visit period as a factor, identity link function and exchangeable within subject working correlation matrix; LS Mean = -82.73, 95% CI 2-sided [-105.00 to -60.46], Standard Error of Mean 11.363
Statistical Analysis 2: Comparison: UX007 (Triheptanoin); Month 4-6; Test type: Superiority; p = 0.0006, GEE model — [p-value comment as in outcome 2, analysis 1]; LS mean = -54.91, 95% CI 2-sided [-86.46 to -23.36], Standard Error of Mean 16.097
Statistical Analysis 3: Comparison: UX007 (Triheptanoin); Month 7-9; Test type: Superiority; p = 0.0019, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean = -52.53, 95% CI 2-sided [-85.62 to -19.45], Standard Error of Mean 16.882
Statistical Analysis 4: Comparison: UX007 (Triheptanoin); Month 10-12; Test type: Superiority; p < 0.0001, GEE model — [p-value comment as in outcome 2, analysis 1]; LS Mean = -82.65, 95% CI 2-sided [-113.13 to -52.17], Standard Error of Mean 15.550

3. Secondary Outcome: Change From Baseline Over Time in CNS Total Score
Description: The CNS evaluates measures of neurological function and development delay, and is the sum of scores for the following domains: Weight, Height, Head Circumference, General Medical Exam, Funduscopic Exam, Cranial Nerves, Stance & Gait, Involuntary Movements, Sensation, Cerebellar Function, Muscle Bulk, Tone & Strength, Myotatic Reflexes, Toe Sign, Other Findings. The CNS is only scored when all domains are measured and ranges from 0 (abnormal exam) to 76 (normal exam). Higher scores are associated with higher neurological function.
Time Frame: Baseline (from NCT01993186), Month 0, Month 6, Month 12, Month 24, Month 36
Population: Participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 12
score on a scale
  Change at Month 0: number analyzed (Participants) | 10
  Change at Month 0 | 11.85 (20.331)
  Change at Month 6: number analyzed (Participants) | 7
  Change at Month 6 | 9.36 (18.495)
  Change at Month 12: number analyzed (Participants) | 7
  Change at Month 12 | 13.64 (21.371)
  Change at Month 24: number analyzed (Participants) | 4
  Change at Month 24 | 3.38 (3.092)
  Change at Month 36: number analyzed (Participants) | 1
  Change at Month 36 | 0.00 (NA) — 1 participant assessed

4. Secondary Outcome: Change From Baseline Over Time in SF-10 Health Survey for Children Physical Summary Score
Description: The SF-10 Health Survey for Children was administered to caregivers of participants aged 5-17 years. Responses are used to generate 2 component summary scores: Physical Summary Score and the Psychosocial Summary Score. The T-score based scale scores were centered so that a score of 50 corresponds to the average score in a comprehensive 2006 sample (a combination of general population and supplemental disability and chronic condition samples). Higher scores are associated with better quality of life.
Time Frame: Baseline (from NCT01993186), Month 0, Month 6, Month 12, Month 18, Month 24, Month 30
Population: Pediatric participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 10
T-score
  Change at Month 0: number analyzed (Participants) | 9
  Change at Month 0 | 0.25 (16.917)
  Change at Month 6: number analyzed (Participants) | 7
  Change at Month 6 | 9.56 (21.522)
  Change at Month 12: number analyzed (Participants) | 6
  Change at Month 12 | -2.67 (9.475)
  Change at Month 18: number analyzed (Participants) | 5
  Change at Month 18 | -9.35 (12.702)
  Change at Month 24: number analyzed (Participants) | 4
  Change at Month 24 | -8.96 (20.075)
  Change at Month 30: number analyzed (Participants) | 2
  Change at Month 30 | 7.74 (2.273)

5. Secondary Outcome: Change From Baseline Over Time in SF-10 Health Survey for Children Psychosocial Summary Score
Description: as for outcome 4
Time Frame: Baseline (from NCT01993186), Month 0, Month 6, Month 12, Month 18, Month 24, Month 30
Population: Pediatric participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 10
T-score
  Change at Month 0: number analyzed (Participants) | 9
  Change at Month 0 | 0.59 (11.049)
  Change at Month 6: number analyzed (Participants) | 7
  Change at Month 6 | -2.29 (12.366)
  Change at Month 12: number analyzed (Participants) | 6
  Change at Month 12 | -7.43 (15.514)
  Change at Month 18: number analyzed (Participants) | 5
  Change at Month 18 | -6.60 (14.987)
  Change at Month 24: number analyzed (Participants) | 4
  Change at Month 24 | -8.25 (15.316)
  Change at Month 30: number analyzed (Participants) | 2
  Change at Month 30 | 8.91 (12.599)

6. Secondary Outcome: Change From Baseline Over Time in SF-12v2 Health Survey PCS Score
Description: SF-12v2 was assessed for adults 18 years of age and older. Eight domain scores were used to generate 2 component summary scores: physical health (PCS) and mental health (MCS). The PCS and MCS scores have mean of 50 and SD of 10. The T-score based scoring method scores the data in relation to U.S. general population T-scores. Therefore, all scores obtained that are below 50 can be interpreted as below the U.S. general population T-score and scores above 50 can be interpreted as above the U.S. general population T-score. Higher global scores are associated with better quality of life.
Time Frame: Baseline (from NCT01993186), Month 0, Month 6, Month 12, Month 18
Population: Adult participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 2
T-score
  Change at Month 0 | 10.25 (5.077)
  Change at Month 6 | 12.37 (5.367)
  Change at Month 12 | 5.09 (1.619)
  Change at Month 18: number analyzed (Participants) | 1
  Change at Month 18 | -0.35 (NA) — 1 participant assessed.

7. Secondary Outcome: Change From Baseline Over Time in SF-12v2 Health Survey MCS Score
Description: as for outcome 6
Time Frame: Baseline (from NCT01993186), Month 0, Month 6, Month 12, Month 18
Population: Adult participants with a baseline and postbaseline assessment at given time point.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | UX007 (Triheptanoin)
Number analyzed (Participants) | 2
T-score
  Change at Month 0 | 8.63 (2.249)
  Change at Month 6 | 5.84 (3.316)
  Change at Month 12 | 6.90 (5.706)
  Change at Month 18: number analyzed (Participants) | 1
  Change at Month 18 | 16.96 (NA) — 1 participant assessed.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 36 months. The mean (SD) treatment duration was 667.9 (357) days.
Arm/Group | UX007 (Triheptanoin)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 13/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX007 (Triheptanoin) (N=15)
Intestinal Obstruction (Gastrointestinal disorders) | 1
Croup Infectious (Infections and infestations) | 1
Ear Infection (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX007 (Triheptanoin) (N=15)
Tachycardia (Cardiac disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 1
Breath Odour (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 1
Thirst (General disorders) | 1
Seasonal Allergy (Immune system disorders) | 1
Ear Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Otitis Media (Infections and infestations) | 1
Otitis Media Acute (Infections and infestations) | 1
Pharyngitis Streptococcal (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Head Injury (Injury, poisoning and procedural complications) | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1
Alanine Aminotransferase Increased (Investigations) | 1
Blood Glucose Increased (Investigations) | 1
Weight Increased (Investigations) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1
Disturbance In Attention (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Head Titubation (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Lethargy (Nervous system disorders) | 3
Petit Mal Epilepsy (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1
Vulvovaginal Pruritus (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1
Hot Flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT02599961/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT02599961/SAP_001.pdf